CLINICAL TRIAL: NCT05702255
Title: Effect of Self- Administered Acupressure on Diarrhea Predominant Irritable Bowel Syndrome Patients' Health Outcomes: a Double Blind- Sham Controlled Randomized Clinical Trial
Brief Title: Self- Administered Acupressure for Diarrhea Predominant Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Maha Gamal Ramadan Asal, Principle investgator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022-9-55
Record Dates: First submitted 2023-01-07; First posted 2023-01-27 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Irritable Bowel Syndrome With Diarrhea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: a randomization sequence will be generated by an independent statistician. The randomization list will be recorded and enclosed in sequentially numbered, opaque envelopes. after finishing baseline assessment, the training researcher will open the envelopes to avoid selection bias. only the training researcher will know the group allocation. Participants and other relevant researchers (the outcome evaluator, data managers, and statisticians) will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active acupoints group (Experimental): All participants in the active group will be treated with basic acupoints Zhongwan (CV 12), Tianshu (ST25) in alternation with Sanyinjiao (SP 6), Zusanli (ST 36). Moreover according to traditional Chinese medicine diagnosis, additional acupoints will be added. The frequency of acupressure treatment will be twice a day for 4 weeks, in total 56 sets.
  Interventions: Other: Active acupressure
- Sham acupoints group (Sham Comparator): All participants on the sham acupoints group will recieive sham Zhongwan (CV 12), sham Tianshu (ST25), sham Sanyinjiao (SP 6), and sham Zusanli (ST 36) acupressure. All the sham points are 2 cm outside and parallel to the actual points which do not match any recognized acupuncture points and are thought to have no therapeutic effect. The frequency of acupressure treatment will be twice a day for 4 weeks, in total 56 sets.
  Interventions: Other: Sham acuptressure

INTERVENTIONS:
Other: Active acupressure — Participants will receive training (2 sessions, 2 days a part) by a training researcher. Patients will be taught on the acupoints location and the acupressure technique. Participants will be verified for the correct location of the acupoints, acupressure technique and strength. Participants will be instructed to use thumb or middle finger to self- press each acupoint using circular movements. The force of pressing must be sufficiently strong but still within a comfortable range. A lubricant will be uses to decrease friction between the acupoints and the finger. Follow up evaluation will be at the end of the week 2 and week 4 .The training researcher will make weekly calls to remind participants to perform acupressure and to answer questions
  Arms: Active acupoints group
Other: Sham acuptressure — The same protocol as the active acupressure group.
  Arms: Sham acupoints group

SUMMARY:
This study aims to assess the effect of active self- administered acupressure compared to sham self- administered acupressure on the health outcome for patient with diarrhea predominant Irritable Bowel Syndrome

DETAILED DESCRIPTION:
Research suggests promising benefits of acupuncture in terms of symptom control and quality of life improvements in patients with irritable bowel syndrome. but the cost of the needle and the invasive nature of the procedure decreases patient compliance with acupuncture. in this respect, acupressure can be taught to patients to allow them to perform it themselves, instead of being administered by practitioners. Self-administered acupressure is less time-intensive, low-cost, and flexible to perform. Nurses involved in irritable bowel syndrome patient care play an active role in the practitioner-patient relationship By assessing the specific symptoms that are present, determining the severity of symptoms and the impact on the irritable bowel syndrome patient's life, and being knowledgeable of available treatment options, the nurse involved in irritable bowel syndrome care becomes an essential conduit of information and a valuable facilitator of a positive practitioner-patient therapeutic relationship. In this way, nurses can help to limit the negative consequences of this common disorder and improve overall treatment outcomes in this population. . Thus this study will be conducted to assess the effectiveness of active self-administered acupressure on diarrhea-predominant irritable bowel syndrome

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diarrhea irritable bowel syndrome symptoms following Rome IV diagnostic criteria
* Agreed to be on a fixed dose of the pharmacological therapy throughout the study

Exclusion Criteria:

* Patients with severe lesions in major organs such as the heart, liver, and kidney, hematopoietic diseases, or tumors
* Eating disorders
* History of major abdominal surgery
* History of neurological and mental illness
* Usage of other treatment rather than the medical treatment regularly 2 weeks before randomization and throughout the study
* Previous history of drug or alcohol abuse 6 months before randomization
* Pregnant and lactating women.
* Patient reporting of adequate relief of their irritable bowel syndrome symptoms the week preceding the randomization
* Patient has too mild symptoms ( obtaining less than 75 on Irritable bowel syndrome symptoms severity scale at the baseline assessment)
* Currently participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Baseline mean of irritable Bowel Syndrome Symptom Severity Score | Immediately before assigning the participants to the study groups
  It is five item questionnaire measuring frequency and intensity of abdominal pain, the severity of abdominal distension, dissatisfaction with bowel habits, and the interference of IBS with daily life. Subjects respond to each question on a 100-point visual analogue scale. The total score ranges from 0 to 500. Subjects can be categorized as having mild (75-175), moderate (175-300), or severe (>300) disease
Change from the baseline irritable Bowel Syndrome Symptom Severity Score at 2 weeks | after 2 weeks from the baseline
  t is five item questionnaire measuring frequency and intensity of abdominal pain, the severity of abdominal distension, dissatisfaction with bowel habits, and the interference of IBS with daily life. Subjects respond to each question on a 100-point visual analogue scale. The total score ranges from 0 to 500. Subjects can be categorized as having mild (75-175), moderate (175-300), or severe (>300) disease
Change from the baseline irritable Bowel Syndrome Symptom Severity Score at 4 weeks | after 4 weeks from the baseline
  t is five item questionnaire measuring frequency and intensity of abdominal pain, the severity of abdominal distension, dissatisfaction with bowel habits, and the interference of IBS with daily life. Subjects respond to each question on a 100-point visual analogue scale. The total score ranges from 0 to 500. Subjects can be categorized as having mild (75-175), moderate (175-300), or severe (>300) disease
Irritable Bowel Syndrome Adequate Relief question | At the baseline
  It is a dichotomous single item that asks participants "Over the past week have you had adequate relief of your irritable Bowel Syndrome symptoms?" . A responder was defined as a patient who answered this question affirmatively.
Irritable Bowel Syndrome Adequate Relief question | After 2 weeks from the baseline
  It is a dichotomous single item that asks participants "Over the past week have you had adequate relief of your irritable Bowel Syndrome symptoms?" . A responder was defined as a patient who answered this question affirmatively.
Irritable Bowel Syndrome Adequate Relief question | After 4 weeks from the baseline
  It is a dichotomous single item that asks participants "Over the past week have you had adequate relief of your irritable Bowel Syndrome symptoms?" . A responder was defined as a patient who answered this question affirmatively.
Mean stool frequency after 2 weeks | After 2 weeks from the patient endorsement
  Defined by the bi-weekly change of frequency of defecation,patient will report the number of defecation per day to calculate it.
Mean change of stool frequency after 4 weeks | After 4 weeks from the patient endorsement
  Defined by the bi-weekly change of frequency of defecation,patient will report the number of defecation per day to calculate it.
Stool consistency | at the baseline
  Defined by the Bristol Stool Form Scale, It is an ordinal scale of stool types ranging from the hardest (Type 1) to the softest (Type 7). Types 1 and2 are considered to be abnormally hard stools while Types 6 and 7 are considered abnormally loose/liquid stools. Type 3, 4 and 5 are considered to be the most normal stool type
Change in the frequency of stool consistency at 2 weeks from the baseline | after 2 weeks from baseline
  defined by the Bristol Stool Form Scale
Change in the frequency of stool consistency at 4 weeks from the baseline | after 4 weeks
  Defined by the Bristol Stool Form Scale, It is an ordinal scale of stool types ranging from the hardest (Type 1) to the softest (Type 7). Types 1 and2 are considered to be abnormally hard stools while Types 6 and 7 are considered abnormally loose/liquid stools. Type 3, 4 and 5 are considered to be the most normal stool type

SECONDARY OUTCOMES:
Demographic and clinical data | before assignment of the participants to the study groups
  A questionnaire will be developed to collect data about participants' age, gender, body mass index, physical activity status, diet, smoking status, medication used.
the baseline mean of psychological distress measured by the Hospital Anxiety and Depression Scale | at the baseline
  the scale contains 14 items, seven statements on each sub-scale which assess symptoms experienced during the past week on four-point rating scale (0 to 3); a higher score depicts a worse condition. For each sub-scale the maximum score is 21. A score of ≥11 is considered a clinically significant disorder, whereas a score between 8 and 10 suggests a mild disorder
Change from the baseline mean of the psychological distress measured by the Hospital Anxiety and Depression Scale at 4 weeks | after 4 weeks from the baseline
  the scale contains 14 items, seven statements on each sub-scale which assess symptoms experienced during the past week on four-point rating scale (0 to 3); a higher score depicts a worse condition. For each sub-scale the maximum score is 21. A score of ≥11 is considered a clinically significant disorder, whereas a score between 8 and 10 suggests a mild disorder
Baseline mean of the quality of Life | at the baseline
  it will be measured by the irritable bowel syndrome quality of Life questionnaire. It consists of 34 items that assess the degree to which irritable bowel syndrome disturbed quality of life for a subject over the past 30 days through eight sub-scales. Each item is rated on a 5-point scale ranging from 1 to 5 with higher values indicating a lower quality of life.
Change from the baseline mean of the quality of life at 4 weeks | Four weeks after the baseline assessment
  it will be measured by the irritable bowel syndrome quality of Life questionnaire. It consists of 34 items that assess the degree to which irritable bowel syndrome disturbed quality of life for a subject over the past 30 days through eight sub-scales. Each item is rated on a 5-point scale ranging from 1 to 5 with higher values indicating a lower quality of life.
Related adverse Events | from the patients endorsement till one week after study completion
  An unfavorable change in the health of a participants that happens during a clinical study or within a week after the study has ended. This change may or may not be caused by the acupressure.
Adherence to the to active and sham self-administered acupressure of the study. | throughout study completion, an average of 4 months
  The adherence will be calculated as percentage of planned sessions of acupressure, and adherence rate above 80% was set as a minimum requirement to be regarded as acceptable
use of rescue medicine | throughout study completion, an average of 4 months
  participants will be asked to report the use of rescue medicine for diarrhea or gastrointestinal symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Maha G Asal, Phd, Principal Investigator — Alexandria University; Zahraa H Ramzy, Phd, Principal Investigator — Alexandria University; Rasha F Ahmed, Phd, Principal Investigator — Alexandria University
Locations (1):
- outpatient clinics of Main University Hospital, Alexandria, Egypt

REFERENCES:
- [Derived] Asal MGR, El-Sayed AAI, Alsenany SA, Ramzy ZH, Dawood RFA. Self-administered active versus sham acupressure for diarrhea predominant irritable bowel syndrome: a nurse-led randomized clinical trial. BMC Nurs. 2025 Jan 28;24(1):106. doi: 10.1186/s12912-024-02594-5. PMID 39875940